CLINICAL TRIAL: NCT01405027
Title: Boceprevir in Community Practice: Assessing Safety, Efficacy, Compliance and Quality of Life, Impact of an Education Program
Brief Title: Impact of Physician Directed Education on Patient Compliance With Hepatitis C Therapy
Acronym: OPTIMAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chronic Liver Disease Foundation (Other)
Collaborators: SCRI Development Innovations, LLC (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDF-MER-001-00; 20111013 (Other: Western Institutional Review Board)
Record Dates: First submitted 2011-07-25; First posted 2011-07-29 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Hepatitis C; Genotype 1
Keywords: HCV; Genotype1; Naive; Partial responder; Relapser
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Early Intervention, Educational; peginterferon alfa-2b; peginterferon alfa-2a; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Ribavirin; Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A - HCEE (Other): Group A - CLDF Hepatology Centers of Educational Expertise (HCEE) are hepatologists experienced in educating health professionals about current developments in the management of chronic liver disease and with clinical trial experience using an HCV protease inhibitor. HCEE investigators provided patient education and management skills training during four (4) educational interventions to Community Site investigators.
  Interventions: Other: Patient education and management skills training
- Group B - Community Sites (Other): Group B - community physicians treating HCV but without clinical trial experience with an HCV protease inhibitor received patient education and management skills training from Hepatology Centers of Educational Expertise (HCEEs) during four (4) educational interventions.
  Interventions: Procedure: Educational Intervention

INTERVENTIONS:
Procedure: Educational Intervention — Receive patient education and management skills training from Hepatology Centers of Educational Expertise (HCEE) during four (4) educational interventions.The CLDF (Sponsor) intends to evaluate the effectiveness of the HCEE led educational interventions in improving a community site's HCV therapeutic management skills and patient outcomes.
  Other Names: Peg-Intron; Pegasys; Victrelis; Pegylated interferon alfa 2B; Pegylated interferon alfa 2A; Boceprevir; Ribavirin
  Arms: Group B - Community Sites
Other: Patient education and management skills training — Community sites received patient education and management skills training by HCEE investigators during four (4) educational interventions.The CLDF (Sponsor) intends to evaluate the effectiveness of the HCEE led educational interventions in improving a community site's HCV therapeutic management skills and patient outcomes.
  Other Names: Peg-Intron; Pegasys; Victrelis; Pegylated interferon alfa 2B; Pegylated interferon alfa 2A; Boceprevir; Ribavirin
  Arms: Group A - HCEE

SUMMARY:
The purpose of this study is to evaluate the impact of a physician directed education program on treatment compliance of hepatitis C patients administered triple drug therapy of pegylated interferon, ribavirin and boceprevir.

DETAILED DESCRIPTION:
The new treatment paradigm for HCV in the era of protease inhibitors will add a level of complexity that was previously not seen with pegylated interferon and ribavirin. In addition to new concepts such as utilization of a lead-in period, compliance with a TID dosing regimen of a third agent, development of resistance, and futility rules and decision points have yet to be assessed in a real life practice setting. The OPTIMAL trial is designed to evaluate the impact of an education program for community sites participating in a CLDF study treating chronic HCV genotype 1 patients. Group A will be comprised of approximately 30 CLDF designated Hepatology Centers of Educational Expertise (HCEE) and Group B will be comprised of approximately 60 community sites. Group A will also deliver the educational program regarding the use of HCV protease inhibitors, and the overall treatment of HCV to approximately two (2) community sites in it's geographic region. Group B will be comprised of community sites that have no previous clinical trial experience with boceprevir or an HCV protease inhibitor. For the purpose of this study, each community site in Group B will be assigned to an HCEE.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hepatitis C (HCV) genotype 1
* Detectable HCV-RNA within 180 days of screening
* Age ≥ 18 years
* Weight > 40 kg
* Patient and partner(s) must agree to use acceptable methods of contraception
* Written informed consent

Exclusion Criteria:

* Known co-infection with HIV or HBV
* Previous interferon or ribavirin regimen requiring discontinuation for an adverse event considered related to ribavirin and/or interferon
* Currently taking or planning on taking any prohibited medications
* Evidence of decompensated liver disease including the presence of clinical ascites, bleeding varices, or hepatic encephalopathy
* Diabetes and/or hypertension with clinically significant ocular examination findings
* Pre-existing psychiatric condition(s)
* History of severe and uncontrolled psychiatric disorders
* Active alcohol or drug abuse (not including marijuana)
* Pre-existing medical condition that could interfere with the patient's participation in the study
* Chronic obstructive pulmonary disease
* Abnormal lab values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2011-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Poordad, MD, Principal Investigator — Chronic Liver Disease Foundation
Locations (43):
- United States (43):
  - California Liver Institute, Beverly Hills, California
  - Samuel Burstein, MD, Calabasas, California
  - William Katkov, MD, Santa Monica, California
  - Sutha Sachar, MD, Torrance, California
  - Harbor UCLA Medical Professional Group, Torrance, California
  - Associates in Gastroenterology, Colorado Springs, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Bay Area Gastroenterology, Clearwater, Florida
  - Digestive Medicine Associates, Hialeah, Florida
  - James Johnson, MD, Lakeland, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - Marwan Iskandarani, MD, North Miami Beach, Florida
  - Advanced Gastro and Liver Disease, Pinellas Park, Florida
  - Lee S. Mitchel, MD, Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - Digestive Disease Consultants, Bourbonnais, Illinois
  - Indiana University, Indianapolis, Indiana
  - Consultants in Gastroenerology, Munster, Indiana
  - Consultants in Gastroenterology, Munster, Indiana
  - Wabash Valley Infectious Disease, Terre Haute, Indiana
  - University of Iowa Health Center, Iowa City, Iowa
  - Metropolitan Gastroenterology Associates, Metairie, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - South Oakland Gastroenterology, Farmington Hills, Michigan
  - Union Lake Clinic, Madison Heights, Michigan
  - GI Medicine Associates, Saint Clair Shores, Michigan
  - Saint Luke's Health Center, Kansas City, Missouri
  - Saint Luke's Hospital, Kansas City, Missouri
  - Michael Fedotin, MD, Kansas City, Missouri
  - St. Louis University Liver Center, St Louis, Missouri
  - Mercy Digestive Disease, St Louis, Missouri
  - North Shore Gastroenterology Associates, Great Neck, New York
  - North Shore University Hospital, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - NY Associates in Gastroenterology, The Bronx, New York
  - Temple Physicians, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Dr. Glenn S. Freed, DO, Pottsville, Pennsylvania
  - Main Line Gastroenterology, Wynnewood, Pennsylvania
  - Gastroenterology Consultants, Live Oak, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Medical Associates of Central Virginia, Lynchburg, Virginia

REFERENCES:
- [Derived] Poordad F, Rustgi V, Brown RS Jr, Patel V, Kugelmas M, Regenstein F, Balart L, LaBrecque D, Brown K, Avila M, Biederman M, Freed G, Smith R, Bernstein M, Arnold H, Cahan J, Fink S, Katkov W, Massoumi H, Harrison S. The impact of an educational program on HCV patient outcomes using boceprevir in community practices (OPTIMAL trial). Therap Adv Gastroenterol. 2015 Sep;8(5):263-9. doi: 10.1177/1756283X15588876. PMID 26327916
- See also: Click here for more information about the Chronic Liver Disease Foundation and Hepatology Centers of Educational Expertise — http://www.chronicliverdisease.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - HCEE: Group A - CLDF Hepatology Centers of Educational Expertise (HCEE) are hepatologists experienced in educating health professionals about current developments in the management of chronic liver disease and with clinical trial experience using an HCV protease inhibitor.
  No Intervention: Deliver patient education and management skills training to community sites during four (4) educational interventions.The CLDF (Sponsor) intends to evaluate the effectiveness of the HCEE led educational interventions in improving a community site's HCV therapeutic management skills and patient outcomes.
- Group B - Community Sites: Group B - community physicians treating HCV but no clinical trial experience with an HCV protease inhibitor
  Educational Intervention: Receive patient education and management skills training from Hepatology Centers of Educational Expertise (HCEE) during four (4) educational interventions.The CLDF (Sponsor) intends to evaluate the effectiveness of the HCEE led educational interventions in improving a community site's HCV therapeutic management skills and patient outcomes.
Period: Overall Study
Arm/Group | Group A - HCEE | Group B - Community Sites
Started | 84 | 113
Completed | 52 | 62
Not Completed | 32 | 51
Not completed — Withdrawn consent | 3 | 0
Not completed — Lost to Follow-up | 16 | 24
Not completed — Investigator judgement | 0 | 2
Not completed — Death | 1 | 0
Not completed — Other or Unknown | 12 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - HCEE | Group B - Community Sites | Total
Number analyzed (Participants) | 84 | 113 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (11.37) | 51.7 (11.27) | 52.0 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 64 | 95
  Male | 53 | 49 | 102
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 50 | 75 | 125
  Black/African American | 19 | 23 | 42
  Asian | 3 | 2 | 5
  Latino | 11 | 10 | 21
  Other | 1 | 3 | 4
Patient Status [Number; unit: participants]
  Treatment Naive | 30 | 69 | 99
  Previous Partial Responder | 12 | 5 | 17
  Relapsed | 17 | 22 | 39
  Compensated Cirrhotic | 9 | 8 | 17
  Historic Null Responder | 16 | 9 | 25
Hepatitis C Virus Genotype [Number; unit: participants]
  1a | 62 | 76 | 138
  1b | 22 | 35 | 57
  Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Treatment Duration Compliance Rate
Description: The primary objective will be to define treatment duration compliance rate (calculated as the actual treatment duration in weeks divided by the expected duration in weeks) based on individual patient treatment goals as defined in the OPTIMAL protocol for HCV patients treated with boceprevir, peginterferon and ribavirin for up to 48 weeks. Rates will be reported for HCEEs (Group A) and community sites enrolled in the Program (Group B).
Time Frame: End of treatment up to treatment week 48
Population: Population analyzed represents patients who had a PCR at treatment weeks where expected duration of treatment could have been determined. Subjects who discontinued the study due to Treatment Futility were considered to have 100% treatment duration compliance.
Measure: Mean (95% Confidence Interval); unit: Percentage of compliance
Arm/Group | Group A - HCEE | Group B - Community Sites
Number analyzed (Participants) | 77 | 102
Percentage of compliance | 85.4 [79.7 to 91.2] | 83.8 [78.4 to 89.2]
Statistical Analysis 1: Comparison: Group A - HCEE vs Group B - Community Sites; Test type: Superiority or Other; p = 0.4864, ANOVA

2. Secondary Outcome: Drug Exposure
Description: Total number of patients receiving treatment over specified time intervals.
Time Frame: End of treatment up to treatment week 48
Measure: Number; unit: participants
Arm/Group | Group A - HCEE | Group B - Community Sites
Number analyzed (Participants) | 84 | 113
participants
  Days 1-7 | 84 | 113
  Days 8-14 | 84 | 112
  Days 15-28 | 83 | 110
  Days 29-56 | 81 | 108
  Days 57-84 | 78 | 100
  Days 85-168 | 73 | 91
  Days 169-252 | 49 | 75
  Days >252 | 26 | 30

3. Secondary Outcome: Determination of the Rate of Sustained Viral Response (SVR) for HCV Patients Treated With Boceprevir, Peginterferon and Ribavirin at Community Sites and at HCEEs.
Description: Rate of SVR was defined as the percentage of participants with HCV-RNA undetectable at follow-up Week 24. All percentages were based on the total number of participants originally randomized/enrolled to that particular arm.
Time Frame: Follow-up week 24
Population: Follow-up SVR includes data collected 10 weeks or greater from last treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Group A - HCEE | Group B - Community Sites
Number analyzed (Participants) | 84 | 113
percentage of participants
  Negative (percent) | 48.8 | 46.0
  Positive (percent) | 23.8 | 26.5
  Missing (percent) | 27.4 | 27.4

4. Secondary Outcome: Short Form Health Survey Measuring Quality of Life Reported at Baseline, End of Treatment, and Follow-up Week 24 (36 Multiple Choice Questions)
Description: Determination of the quality of life for HCV patients treated with boceprevir, peginterferon and ribavirin at community sites and at HCEEs.
  Patient scores per subscale (8) were obtained by subtracting the lowest possible raw score from the actual raw score x 100, divided by the lowest possible raw score subtracted from the highest possible raw score. Subscale scores were averaged (with standard deviation) for Group A and Group B. Composite Scores are standardized to the general US population having a mean of 50 and a standard deviation of 10. Higher score = improved quality of life.
Time Frame: Baseline, end of treatment, follow-up week 24
Population: The Quality of Life scores are derived from the responses from subjects who completed questionnaires at protocol-scheduled timepoints.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Group A - HCEE | Group B - Community Sites
Number analyzed (Participants) | 77 | 109
score
  Physical Component Score - baseline | 44.6 (12.58) | 45.5 (11.80)
  Physical Component Score - End of treatment | 42.9 (10.38) | 43.7 (9.21)
  Physical Component Score - Follow-up week | 49.2 (8.75) | 49.4 (11.34)
  Mental Component Score - Baseline | 52.2 (8.78) | 51.4 (9.08)
  Mental Component Score - End of treatment | 45.3 (10.68) | 45.2 (10.05)
  Mental Component Score - Follow-up week | 54.8 (8.49) | 51.9 (8.44)
  Physical Functioning - Baseline | 76.1 (29.27) | 77.1 (26.23)
  Physical Functioning - End of treatment | 68.3 (26.45) | 70.3 (24.00)
  Physical Functioning - Follow-up week | 84.2 (24.35) | 82.3 (24.19)
  Physical Role Functioning - Baseline | 71.0 (40.16) | 68.0 (41.22)
  Physical Role Functioning - End of treatment | 47.1 (42.96) | 47.0 (42.76)
  Physical Role Functioning - Follow-up week | 80.7 (31.38) | 81.8 (33.67)
  Bodily Pain - Baseline | 63.1 (29.62) | 68.9 (29.02)
  Bodily Pain - End of treatment | 65.1 (24.89) | 66.0 (22.04)
  Bodily Pain - Follow-up week | 76.7 (24.33) | 73.8 (27.60)
  General Health - Baseline | 67.7 (21.44) | 65.7 (23.42)
  General Health - End of treatment | 65.9 (21.93) | 69.0 (20.05)
  General Health - Follow-up week | 74.6 (18.28) | 74.0 (19.24)
  Vitality - Baseline | 57.5 (23.75) | 58.2 (23.12)
  Vitality - End of treatment | 44.6 (25.55) | 43.0 (23.61)
  Vitality - Follow-up week | 71.7 (20.37) | 65.7 (18.86)
  Social Functioning - Baseline | 82.4 (24.21) | 82.8 (24.70)
  Social Functioning - End of treatment | 66.0 (26.35) | 67.9 (25.86)
  Social Functioning - Follow-up week | 89.8 (16.89) | 87.2 (18.04)
  Emotional Role Functioning - Baseline | 86.6 (28.75) | 80.3 (34.18)
  Emotional Role Functioning - End of treatment | 61.1 (42.15) | 64.2 (42.76)
  Emotional Role Functioning - Follow-up week | 85.6 (31.66) | 82.0 (32.01)
  Mental Health - Baseline | 76.4 (16.89) | 76.6 (18.45)
  Mental Health - End of treatment | 69.5 (19.61) | 68.5 (17.36)
  Mental Health - Follow-up week | 83.3 (15.34) | 77.2 (15.74)

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Description of the adverse events and rate of events of boceprevir, peginterferon and ribavirin in HCV patients treated at community sites and at HCEEs
Time Frame: Throughout entire study, at end of treatment and follow up week 24
Measure: Number; unit: participants
Arm/Group | Group A - HCEE | Group B - Community Sites
Number analyzed (Participants) | 84 | 113
participants | 77 | 95

ADVERSE EVENTS:
Arm/Group | Group A - HCEE | Group B - Community Sites
Serious Adverse Events (participants affected / at risk) | 6/84 | 8/113
Other Adverse Events (participants affected / at risk) | 77/84 | 92/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - HCEE (N=84) | Group B - Community Sites (N=113)
Fatigue (General disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Stroke (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - HCEE (N=84) | Group B - Community Sites (N=113)
Fatigue (General disorders) | 54 | 28
Irritability (General disorders) | 12 | 3
Influenza like Illness (General disorders) | 10 | 2
Pyrexia (General disorders) | 10 | 3
Malaise (General disorders) | 2 | 9
Nausea (Gastrointestinal disorders) | 36 | 25
Diarrhoea (Gastrointestinal disorders) | 20 | 15
Vomiting (Gastrointestinal disorders) | 9 | 7
Constipation (Gastrointestinal disorders) | 5 | 10
Stomatitis (Gastrointestinal disorders) | 5 | 5
Anaemia (Blood and lymphatic system disorders) | 42 | 44
Neutropenia (Blood and lymphatic system disorders) | 18 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 17
Headache (Nervous system disorders) | 22 | 17
Dysgeusia (Nervous system disorders) | 16 | 17
Dizziness (Nervous system disorders) | 11 | 9
Rash (Skin and subcutaneous tissue disorders) | 24 | 27
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Insomnia (Psychiatric disorders) | 19 | 16
Depression (Psychiatric disorders) | 15 | 11
Anxiety (Psychiatric disorders) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 12
Decreased appetite (Metabolism and nutrition disorders) | 11 | 10
Weight decreased (Investigations) | 4 | 7
Hypothyroidism (Endocrine disorders) | 3 | 7

LIMITATIONS AND CAVEATS:
Smaller sample size than expected due to changing treatment landscape for HCV during course of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less